CLINICAL TRIAL: NCT00619099
Title: Randomized Open-label Phase 2 Study of Low Dose Dacogen® for Injection (Decitabine) in Patients With Low or Intermediate 1 Risk Myelodysplastic Syndromes
Brief Title: A Study of Decitabine Given Subcutaneously to Adults With Low or Intermediate-1 Risk Myelodysplastic Syndromes (MDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DACO-026
Record Dates: First submitted 2008-02-08; First posted 2008-02-20 (Estimated); Results first posted 2013-09-18 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-09

CONDITIONS: Myelodysplastic Syndrome
Keywords: Myelodysplastic Syndrome; Decitabine; Dacogen; MGI PHARMA, Inc.
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: decitabine
- 2 (Experimental)
  Interventions: Drug: decitabine

INTERVENTIONS:
Drug: decitabine — Schedule A: decitabine will be administered subcutaneously (SQ) daily for 3 consecutive days (Days 1 to 3) every 28 days. The dose will be 20 mg/m^2/day. One course will be considered 28 days.
  Other Names: Dacogen
  Arms: 1
Drug: decitabine — Schedule B: decitabine will be administered SQ every 7 days for 21 days (Days 1, 8, and 15) followed by 7 days without an administration of decitabine. The dose will be 20 mg/m^2/day. One course will be considered 28 days.
  Other Names: Dacogen
  Arms: 2

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of two different dose schedules of DACOGEN® (decitabine) for Injection in patients with Myelodysplastic Syndromes (MDS).

DETAILED DESCRIPTION:
This is a randomized open-label Phase 2 efficacy and safety study of two (2) subcutaneous (SQ) dosing schedules of decitabine in subjects with Low or Intermediate 1 Risk MDS. This study will be conducted in up to 6 study centers in the United States.

The primary efficacy outcome is the overall improvement rate. These two doses will be administered subcutaneously. The probability that one schedule is superior to the other will be estimated, and the level of toxicity for each schedule will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet the following criteria to be enrolled in this study:

1. Male or female patients age 18 years and older.
2. Patients must sign an institutional review board (IRB)-approved informed consent form, and understand the investigational nature of this study and its potential hazards prior to initiation of any study-specific procedures or treatment.
3. Must have Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
4. Adequate renal and hepatic function (creatinine < 2 times upper limit of normal, total bilirubin of < 2 times upper limit of normal, and AST and ALT ≤ 2 times upper limit of normal) unless proven to be related to disease infiltration.
5. Female patients need a negative serum or urine pregnancy test within 7 days prior to study drug administration (applies only if patient is of childbearing potential. Non-childbearing is defined as ≥ 1 year postmenopausal or surgically sterilized).
6. Women of childbearing potential and men must use contraception. Men and women must continue birth control for the duration of the study.
7. Patients with Low or Intermediate-1 Risk MDS by the International Prognostic Scoring System (IPSS) classification.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study:

1. Women who are pregnant or nursing.
2. Those who have received prior therapy with decitabine.
3. Prior therapy with azacitidine (Vidaza®).
4. Those who received growth factor support or lenalidomide in the 30 days prior to the first dose of decitabine.
5. Those who have received an investigational agent 30 days prior to the first dose of decitabine.
6. Patients with active, uncontrolled, systemic infection considered opportunistic, life threatening or clinically significant; or any severe, concurrent disease, which, in the judgment of the Investigator and after discussion with the Sponsor and Primary Investigator, would make the patient inappropriate for study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2008-05; Primary Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Gabrail Cancer Center, Canton, Ohio
  - Landmark Medical Center, Woonsocket, Rhode Island
  - Sarah Cannon Research, Nashville, Tennessee
  - M. D. Anderson, Houston, Texas

REFERENCES:
- [Derived] Garcia-Manero G, Jabbour E, Borthakur G, Faderl S, Estrov Z, Yang H, Maddipoti S, Godley LA, Gabrail N, Berdeja JG, Nadeem A, Kassalow L, Kantarjian H. Randomized open-label phase II study of decitabine in patients with low- or intermediate-risk myelodysplastic syndromes. J Clin Oncol. 2013 Jul 10;31(20):2548-53. doi: 10.1200/JCO.2012.44.6823. Epub 2013 Jun 3. PMID 23733767

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 5 centers in U.S. during the period of Jun 2008 to Aug 2011.
Groups:
- Schedule A: SQ 3 Consecutive Days: Decitabine : Schedule A: decitabine will be administered subcutaneously (SQ) daily for 3 consecutive days (Days 1 to 3) every 28 days. The dose will be 20 mg/m^2/day. One course will be considered 28 days.
- Schedule B: SQ Once Every 7 Days: Decitabine : Schedule B: decitabine will be administered SQ every 7 days for 21 days (Days 1, 8, and 15) followed by 7 days without an administration of decitabine. The dose will be 20 mg/m^2/day. One course will be considered 28 days.
Period: Overall Study
Arm/Group | Schedule A: SQ 3 Consecutive Days | Schedule B: SQ Once Every 7 Days
Started | 44 (All randomized subjects) | 23 (All randomized subjects)
Received at Least 2 Cycles of Treatment | 43 (Subjects included in the Modified Intent to Treat Population) | 22 (Subjects included in the Modified Intent to Treat Population)
Completed | 11 | 4
Not Completed | 33 | 19
Not completed — Progressive Disease | 7 | 5
Not completed — Allogeneic Bone Marrow Transplantation | 2 | 1
Not completed — Adverse Event | 4 | 3
Not completed — Emergence of Clinically Significant Lab | 1 | 2
Not completed — Withdrawal by Subject | 10 | 2
Not completed — Physician Decision | 9 | 6

BASELINE CHARACTERISTICS:
Population: Modified Intent to Treat (mITT) Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Schedule A: SQ 3 Consecutive Days | Schedule B: SQ Once Every 7 Days | Total
Number analyzed (Participants) | 43 | 22 | 65
Age Continuous [Mean (Standard Deviation); unit: years] | 66.9 (14.39) | 70.5 (9.86) | 68.2 (13.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 2 | 20
  Male | 25 | 20 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 42 | 20 | 62
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 0 | 5
  White | 35 | 20 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: The Overall Improvement Rate
Description: Defined as proportion of patients having complete remission (CR), partial remission (PR), marrow complete remission (mCR), or hematologic improvement.
  Based on Modified International Working Group Response Criteria for Altering Natural History of Myelodysplastic Syndromes.
  Complete Remission: Bone marrow: ≤ 5% myeloblasts with normal maturation of all cell lines. Persistent dysplasia will be noted. Peripheral blood Hgb ≥ 11 g/dL; Platelets ≥ 100 X 109/L; Neutrophils ≥ 1.0 X 109/Lb; Blasts 0%.
  Partial Remission: All CR criteria if abnormal before treatment except: Bone marrow blasts decreased by ≥ 50% over pretreatment but still > 5%.
  Marrow Complete Remission: Bone marrow: ≤ 5% myeloblasts and decrease by ≥ 50% over pretreatment. Peripheral blood: if hematological improvement responses, they will be noted in addition to marrow CR.
  HI Improvement: shown in increases in hemoglobin, platelet and neutrophil response.
Time Frame: Up to one year
Population: Modified Intent to Treat (mITT) Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Schedule A: SQ 3 Consecutive Days | Schedule B: SQ Once Every 7 Days
Number analyzed (Participants) | 43 | 22
Percentage of Participants
  Overall Improvement Rate | 23.3 | 22.7
  Complete Response | 16.3 | 0
  Marrow Complete Response | 0 | 4.5
  Partial Response | 0 | 4.5
  Hematologic Improvement | 7.0 | 13.6

ADVERSE EVENTS:
Arm/Group | Schedule A: SQ 3 Consecutive Days | Schedule B: SQ Once Every 7 Days
Serious Adverse Events (participants affected / at risk) | 18/43 | 10/22
Other Adverse Events (participants affected / at risk) | 43/43 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Schedule A: SQ 3 Consecutive Days (N=43) | Schedule B: SQ Once Every 7 Days (N=22)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 1
Streptococcal bacteremia (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Neutropenia sepsis (Infections and infestations) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 2
Infection worsening (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Pneumonitis (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Escherichia bacteremia (Infections and infestations) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Conjunctival hemorrhage (Eye disorders) | 1 | 0
Retinal hemorrhage (Eye disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Bladder obstruction (Renal and urinary disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Myelodysplastic syndrome worsening (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute myeloid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cerebral hemorrhage (Nervous system disorders) | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Subdural hematoma (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Stem cell transplant (Surgical and medical procedures) | 1 | 0
Aortic Aneurysm (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Schedule A: SQ 3 Consecutive Days (N=43) | Schedule B: SQ Once Every 7 Days (N=22)
Anemia (Blood and lymphatic system disorders) | 24 | 9
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0
Leukopenia (Blood and lymphatic system disorders) | 18 | 10
Neutropenia (Blood and lymphatic system disorders) | 27 | 15
Thrombocytopenia (Blood and lymphatic system disorders) | 18 | 12
Vision blurred (Eye disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Constipation (Gastrointestinal disorders) | 6 | 6
Diarrhea (Gastrointestinal disorders) | 7 | 6
Hematochezia (Gastrointestinal disorders) | 0 | 2
Hemorrhoids (Gastrointestinal disorders) | 0 | 2
Mouth hemorrhage (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 12 | 3
Oral pain (Gastrointestinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 4 | 2
Asthenia (General disorders) | 5 | 2
Chills (General disorders) | 4 | 0
Edema peripheral (General disorders) | 7 | 5
Fatigue (General disorders) | 17 | 10
Injection site pain (General disorders) | 7 | 4
Injection site reaction (General disorders) | 1 | 2
Pyrexia (General disorders) | 14 | 6
Hyperbilirubinemia (Hepatobiliary disorders) | 3 | 1
Cellulitis (Infections and infestations) | 2 | 2
Nasopharyngitis (Infections and infestations) | 3 | 1
Pneumonia (Infections and infestations) | 3 | 3
Sinusitis (Infections and infestations) | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 3
Urinary tract infection (Infections and infestations) | 7 | 1
Contusion (Injury, poisoning and procedural complications) | 6 | 4
Fall (Injury, poisoning and procedural complications) | 3 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 2
Transfusion reaction (Injury, poisoning and procedural complications) | 3 | 0
Alanine aminotransferase increased (Investigations) | 4 | 1
Aspartate aminotransferase increased (Investigations) | 5 | 2
Blood creatinine increased (Investigations) | 4 | 4
Blood urea increased (Investigations) | 2 | 4
Cardiac murmur (Investigations) | 5 | 5
Transaminases increased (Investigations) | 0 | 2
Weight decreased (Investigations) | 7 | 5
Weight increased (Investigations) | 2 | 3
Decreaed appetite (Metabolism and nutrition disorders) | 5 | 9
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 10 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 5
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Joint swelling (Musculoskeletal and connective tissue disorders) | 4 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 3
Dizziness (Nervous system disorders) | 11 | 6
Headache (Nervous system disorders) | 8 | 2
Hypoaesthesia (Nervous system disorders) | 5 | 2
Memory impairment (Nervous system disorders) | 2 | 2
Somnolence (Nervous system disorders) | 3 | 0
Tremor (Nervous system disorders) | 2 | 2
Anxiety (Psychiatric disorders) | 3 | 0
Insomnia (Psychiatric disorders) | 5 | 3
Hematuria (Renal and urinary disorders) | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 3
Erythema (Skin and subcutaneous tissue disorders) | 3 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 4
Petechiae (Skin and subcutaneous tissue disorders) | 3 | 3
Pruritis (Skin and subcutaneous tissue disorders) | 6 | 3
Rash (Skin and subcutaneous tissue disorders) | 4 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 3
Sinus operation (Surgical and medical procedures) | 4 | 0
Hypertension (Vascular disorders) | 3 | 0
Hypotension (Vascular disorders) | 4 | 3
Orthostatic hypotension (Vascular disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No